CLINICAL TRIAL: NCT02465892
Title: Pillars4Life Randomized Control Trial
Brief Title: Pillars4Life Trial
Acronym: Pillars4Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: Pro00061381
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2016-12

CONDITIONS: Breast Cancer; Lung Cancer; Esophageal Cancer; Colon Cancer; Pancreatic Cancer; Liver Cancer; Renal Cancer; Bladder Cancer; Prostate Cancer; Ovarian Cancer; Cervical Cancer; Uterine Cancer
Keywords: cancer; stress; chronic pain; anxiety; coping; balance; online course; psychosocial; support; tools
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Esophageal Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms; Neoplasms; Chronic Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Subjects in this group will continue receiving standard care from their provider team.
- Pillars4Life (Experimental): Subjects in this group will complete the Pillars4Life online coping skills curriculum.
  Interventions: Behavioral: Pillars4Life

INTERVENTIONS:
Behavioral: Pillars4Life — The Pillars4Life program will guide participants through activities that will help to identify stress and anxiety triggers, plan ways to cope with the stress of life and cancer, manage anxiety, deal with chronic pain, and balance competing priorities in life.
  Arms: Pillars4Life

SUMMARY:
This study aims to explore whether cancer patients can benefit from completing the Pillars4Life online coping program. This randomized control trial will have half its subject completing the program and the other half receiving standard care in order to measure whether the program is beneficial in dealing with stress, anxiety, and particularly chronic pain that often accompany a cancer diagnosis.

DETAILED DESCRIPTION:
Subjects will complete three online surveys as part of the study. Each subject who completes the first survey will be randomized to either the control group who receive standard care from their care team or to complete the 9-week Pillars4Life curriculum. Subjects completing the Pillars4Life program will select a course day/time that works for them from those offered. Each week the program will send an email approximately 15 minutes before class time with a link. Subjects will click the link to go to the "classroom," where they will enter their name and phone number. The program will call the number provided and the subject will listen to the audio over the phone, while watching the guide and activities in the virtual classroom on their computer. Each class will last about an hour.

All subjects will complete two additional surveys, at approximately 9 weeks and 18 weeks after enrolling in the study.

ELIGIBILITY:
Inclusion Criteria:

* Current pain level ≥3 and at least one prior score ≥3 on a 0-10 scale as reported in EPIC;
* Age ≥18 years
* Diagnosed with Breast, GI, GU, GYN, or Thoracic cancer
* Actively receiving care at the Duke Cancer Center, Durham Regional Hospital, or Duke Raleigh Hospital
* Able/willing to have an online interaction with the Pillars4Life online CORE program curriculum
* Life expectancy ≥6 months
* Providing informed consent
* Able to read/write English.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Chronic pain | 9 weeks
  Subjects will report how much chronic pain they have and how they are coping with it.

SECONDARY OUTCOMES:
Stress | 9 weeks
  Subjects will report how much stress they are under they have and how they are coping with it.
Anxiety | 9 weeks
  Subjects will report how much anxiety they have and how they are coping with it.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia K Smith, PhD, MSW, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States